CLINICAL TRIAL: NCT00854139
Title: Combined HLA-matched Bone Marrow and Kidney Transplantation for Multiple Myeloma With Renal Failure
Brief Title: Combined Bone Marrow Transplantation (BMT) and Renal Transplant for Multiple Myeloma (MM) With End Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas Spitzer, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKD01
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma; End Stage Renal Disease
Keywords: Multiple myeloma; Renal failure; Kidney transplant
MeSH Terms: conditions — Multiple Myeloma; Kidney Failure, Chronic; Renal Insufficiency | interventions — Cyclophosphamide; Antilymphocyte Serum; Cyclosporine; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone marrow and renal transplant (Experimental): Cyclophosphamide, anti-thymocyte globulin, thymic irradiation conditioning and kidney transplant and bone marrow transplant from a related donor for patients with multiple myeloma and end stage renal disease with cyclosporine for graft versus host disease prophylaxis
  Interventions: Drug: Cyclophosphamide, anti-thymocyte globulin; Procedure: Kidney transplant; Radiation: Thymic irradiation; Procedure: Bone marrow transplant from a related donor

INTERVENTIONS:
Drug: Cyclophosphamide, anti-thymocyte globulin — Cyclophosphamide 60 mg/kg IV on Day -5, -4 Anti-thymocyte globulin 20 mg/kg IV on Day -1, Day +1, +3, +5
  Cyclosporine starting on Day -1 at 5 mg/kg daily I.V. and reduced to 3 mg/kg on Day +4, and adjusted to provide a trough whole blood concentration of 250-400 ng/mL. The route of administration will be changed to oral as soon as the patient is able to tolerate oral medications
  Other Names: Cyclosporine
Procedure: Kidney transplant — On Day 0 the renal transplant is performed according to standard surgical techniques, preferably using an iliac fossa, extraperitoneal approach
Radiation: Thymic irradiation — Thymic irradiation 7 Gy on Day -1
Procedure: Bone marrow transplant from a related donor — • Donor bone marrow (> 2 x 108 nucleated cells/kg of recipient body weight) is prepared for infusion according to the standard procedure at the medical center. A total of 15,000 Units of heparin is mixed with the marrow, which is infused at a rate of 300-500 cc/hr. The infusion begins in the operating room as soon as the vascular anastomosis of the renal allograft has been completed. Protamine, 25 mg, is administered I.V. after completion of the first half of the bone marrow infusion. If a partial thromboplastin time measured after completion of the marrow infusion is > 60 seconds, the protamine treatment shall be repeated

SUMMARY:
The primary objective is to cure multiple myeloma with less toxic allogeneic bone marrow transplantation while inducing renal allograft tolerance through mixed chimerism in patients with end stage renal failure and multiple myeloma

DETAILED DESCRIPTION:
The induction of transplantation tolerance involves the specific elimination of the immune response to the transplant but not to other antigens. In the realm of kidney transplantation, tolerance means that the recipient is unable to detect the donor transplant kidney as foreign, and therefore the recipient is unable to reject the kidney. Donor bone marrow engraftment leads to kidney graft tolerance in animal models. Renal failure is a major complication of multiple myeloma, a plasma cell malignancy for which the only known cure is allogeneic bone marrow transplantation. Standard bone marrow transplantation is associated with frequent toxicity in patients with multiple myeloma, and is generally no considered an option for those patients with end stage renal disease. Myeloma patients are excluded from conventional renal transplantation protocols because of their underlying malignancy. A less toxic bone marrow transplantation protocol, combined with renal transplantation, could provide an opportunity for cure of the myeloma and correction of ESRD in patients with this disease. In addition, successful marrow engraftment may be expected to lead to a state of tolerance. Successful implementation of tolerance would be a major benefit to transplant recipients. The significance of developing tolerance is that the patient would be spared the disabling complications of indefinite immunosuppression, which include infections, cataracts, osteoporosis, diabetes, atherosclerosis, hypertension, and malignancy

ELIGIBILITY:
Recipient Inclusion Criteria

1. Participants with end-stage renal failure due to or in association with greater than or equal to stage II multiple myeloma
2. Males or females 18 - 65 years of age.
3. Participants must have an HLA-matched or one of six HLA A, B, or DR antigen-mismatched related donor, with high resolution molecular DR allele determination.
4. Men and women of reproductive potential must agree to use a reliable method of birth control during the treatment, and women should do so for a period of 2 years following the transplant.
5. Participants should be on dialysis or have a CrCl <20 ml/min.
6. Participants must receive medical clearance by a cardiologist prior to conditioning for transplant.
7. Life expectancy greater than or equal to 6 months.
8. Recipient ability to understand and provide informed consent.

Recipient Exclusion Criteria:

1. Evidence of active infection as defined by: a) clinical syndrome consistent with viral or bacterial infection (e.g., influenza, URI, UTI) or b) fever with a clinical site of infection identified, or c) microbiologically documented infection, including, but not limited to, bacteremia or septicemia.
2. Participation in other investigational drug use at the time of enrollment.
3. Contraindication to therapy with any one of the proposed agents (e.g., history of allergy to horse serum in ATG).
4. Serologic positivity to HIV, HCV, or HbsAg positivity.
5. Women of childbearing age in whom adequate contraception cannot be maintained.
6. Malignancy within the past two years other than multiple myeloma, excluding basal cell carcinoma of the skin and carcinoma in situ of the cervix.
7. AST/ALT > 3 x normal or bilirubin > 1.5 x normal (unless due to Gilbert's syndrome).
8. Pregnancy or uncontrolled serious medical illness not related to underlying myeloma.
9. Cardiac ejection fraction < 40% by echocardiogram; individual assessment if ejection fraction between 40% and 50%.
10. FEV1 < 50% predicted or corrected DLCO < 50% predicted.
11. ABO blood group incompatibility in the host-vs-graft direction.

Donor Inclusion Criteria:

1. HLA-matched or one of six HLA A, B, or DR antigen-mismatched related male or female donor 18-65 years of age.
2. ECOG performance status 0 or 1.
3. Excellent health per conventional pre-donor history (medical and psychosocial evaluation).
4. Acceptable laboratory parameters (hematology in normal or near-normal range; liver function < 2 times the upper limit of normal and normal creatinine).
5. Compatible ABO blood group.
6. Negative donor lymphocyte crossmatch.
7. No positive testing for viral infection (HbsAg, HIV, HCV, HTLV-1).
8. Cardiac/Pulmonary evaluation within normal limits (CXR, EKG).
9. Donor ability to understand and provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2001-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Remission status of multiple myeloma | 3 years
Renal allograft acceptance and ability to discontinue immunosuppressive therapy | 3 years

SECONDARY OUTCOMES:
Graft versus host disease (GVHD) | 3 years
Opportunistic infections | 3 years
T cell recovery and immune reconstitution | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Spitzer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States